CLINICAL TRIAL: NCT07009353
Title: A PHASE 1, OPEN-LABEL, 2-ARM PARALLEL STUDY TO INVESTIGATE THE ABSORPTION, DISTRIBUTION, METABOLISM AND EXCRETION OF PF-07054894 USING 2 14C-RADIOLABELED PF-07054894 AND TO ASSESS THE ABSOLUTE BIOAVAILABILITY AND FRACTION ABSORBED OF PF-07054894 IN HEALTHY ADULT MALE PARTICIPANTS USING A 14C-MICROTRACER APPROACH
Brief Title: A Study to Learn How the Study Medicine Called [14C]PF-07054894 is Processed by the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C4151008; 2024-519882-23-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-05-05; First posted 2025-06-06 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1 Period 1 and Period 2 (Experimental): Period 1: This is designed to evaluate the metabolic fate and extent of excretion of PF-07054894 following the study drug administration via the intended clinical route of administration (oral) of [cyclobutenyl-14C]PF-07054894. In order to assess the metabolic fate of [14C]PF-07054894, metabolites of [14C]PF-07054894 circulating in plasma and eliminated in urine and feces following oral administration.
  Period 2: This is designed to evaluate oral bioavailability of a drug and also allow to estimate the fraction of the dose absorbed of the oral PF-07054894 dose. Determination of the fraction of the dose absorbed will provide information on the total PF-07054894 dose absorbed, regardless of the fate of that dose after absorption (eg, metabolism, degradation).
  Interventions: Drug: PF-07054894
- Cohort 2 Period 1 (Experimental): This is designed to further evaluate the cleavage of PF-07054894, which was identified in plasma samples from a preliminary investigation of metabolism in the FIH study. The metabolic fate and extent of excretion of PF-07054894 following the study drug administration via the intended clinical route of administration (oral) of - [methyl-14C]PF-07054894 will be evaluated.
  Interventions: Drug: PF-07054894

INTERVENTIONS:
Drug: PF-07054894 — Cohort 1 Period 1 - Oral [cyclobutenyl-14C]PF-07054894 under fasted state. Cohort 1 Period 2: Oral unlabeled PF-07054894 followed by IV [cyclobutenyl-14C]PF-07054894 fusion over approximately 15 minutes at approximately 1.5 hours after the administration of the oral unlabeled dose.
  Cohort 1 Period 2: Oral unlabeled PF-07054894 followed by IV [cyclobutenyl-14C]PF-07054894 fusion over approximately 15 minutes at approximately 1.5 hours after the administration of the oral unlabeled dose.
  Arms: Cohort 1 Period 1 and Period 2
Drug: PF-07054894 — Cohort 2 Period 1 - Oral [Methyl-14C]PF-07054894 under fasted state.
  Arms: Cohort 2 Period 1

SUMMARY:
The purpose of this study is to learn how quickly and to what extent the study medicine (PF-07054894) is absorbed, broken down, and eliminated from the body.

DETAILED DESCRIPTION:
There are two groups in this study:

* Cohort 1 (which has 2 periods)
* Cohort 2 (has 1 period) Participants will only have to participate in one of the 2 Cohorts.
* In Cohort 1 - Period 1, the study will check how the study medicine (PF-07054894) is removed from the body. In Period 2, the study will find out how well the study medicine is absorbed by the body when given by mouth compared to an intravenous route. (solution of the study medicine is injected directly into a vein). For this period, the PF-07054894 that is injected into the vein is radioactively labeled, but the dose given by mouth is not radioactively labeled. Radioactively labelled are compounds where one or more atoms have been replaced with a radioactive element. This allows researchers to track their movement within cells.
* In Cohort 2 - a different radioactive labelled material is used than the one of Cohort 1. This is done to see how PF 07054894 is removed from the body. The study will also look at how safe the study medicine is and how well it is tolerated when it is given to healthy people.

Participants in Cohort 1 will be involved in this study for about 10 weeks and about 8 weeks for those in Cohort 2. Participants in Cohort 1 will stay in the study clinic in Period 1 for up to 15 days (14 nights) and 8 days (7 nights) in Period 2. Participants in Cohort 2 will stay in the study clinic for up to 15 days (14 nights).

For Period 1 of both Cohort 1 and 2, the study doctor will be checking the levels of radioactively labeled study medicine in body frequently from Day 7 onwards in urine, stool, and any vomit and will let participants know as soon as possible if they have to stay longer or if they can go home. The duration of participants' stay will depend on how quickly or slowly the radioactively labeled study compound leaves their body.

For Period 2, participants will have to stay in the study clinic for 8 days (7 nights) and leave the study clinic on Day 7. However, if the study doctor believes it is necessary to protect participant's health, they may be asked to remain in the study clinic after Day 7.

ELIGIBILITY:
1. Healthy male, aged 18 years to 65 years at screening.
2. Body mass index (BMI) of about 18 to 32 kilogram per meter squared, and a total body weight greater than 50 kilograms (110 pounds).
3. Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only Male participants aged 18 years to 65 years inclusive (or the minimum age of consent in accordance with local regulations) at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests.
Enrollment: 10 (Actual)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Cumulative recovery (%) of radioactivity in urine and feces (adjusted for vomitus, if any), expressed as a percent of total oral radioactive dose administered. | Period 1 of Cohort 1 & 2 pre-dose to maximum Day 14
  To characterize the rate and extent of excretion of total radioactivity following administration of a single oral dose of [14C]PF-07054894(Period 1 of Cohort 1 & 2).
Metabolite identification/profiling in feces, plasma and urine | Period 1 of Cohort 1 & 2 pre-dose to maximum Day 14

SECONDARY OUTCOMES:
Cumulative recovery (%) of radioactivity in plasma expressed as a percent of total oral radioactive dose administered. | Period 1 of Cohort 1 & 2 pre-dose to maximum Day 14
Dose normalized AUCinf of intravenous radiolabeled PF-07054894 in plasma (if data permit). | Period 2 Cohort 1 pre-dose to maximum Day 7
  Dose normalized area under the plasma concentration-time profile from time zero extrapolated to infinite time following administration of a single intravenous dose of radiolabeled PF-07054894.
The fraction of PF-07054894 dose absorbed (Fa). | Period 2 Cohort 1 pre-dose to maximum Day 7
  Fa calculated from the ratio of total recovered radioactivity [14C] in urine following single dose administration of [14C]PF-07054894 orally in Period 2 Cohort 1
The absolute oral bioavailability (F) of PF-07054894. | Period 1 of Cohort 1 pre-dose to maximum Day 14 and Period 2 Cohort 1 pre-dose to maximum Day 7
  The ratio of dose-normalized plasma AUCinf of oral PF-07054894 and IV administration of [14C]PF-07054894 in Period 2 (Cohort 1).
Number of participants with treatment emergent clinically significant laboratory abnormalities | From pre-dose to 28 days post-dose for Cohort 1 and Cohort 2
Number of participants with treatment emergent clinically significant abnormal ECG measurements | From pre-dose to 28 days post-dose for Cohort 1 and Cohort 2
Number of participants with treatment emergent clinically significant abnormal vital measurements | From pre-dose to 28 days post-dose for Cohort 1 and Cohort 2
Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) | From pre-dose to 28 days post-dose for Cohort 1 and Cohort 2
Maximum Observed Plasma Concentration (Cmax) of PF-07054894 | Day 1 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240-, 264-, 288- and 312-hours post-dose
Area Under the Curve from Time Zero to Last Quantifiable Concentration (AUClast) of PF-07054894 | Day 1 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240-, 264-, 288- and 312-hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-07054894 | Day 1 pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240-, 264-, 288- and 312-hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4151008